CLINICAL TRIAL: NCT02422394
Title: Eltrombopag for Inherited Thrombocytopenias
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Alessandro Pecci, researcher of Internal Medicine and assistant physician at the Unit of Internal Medicine 3, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Eltrombo-IT-2014
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Inherited Platelet Disorder
MeSH Terms: interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eltrombopag (Experimental): Phase 1: Eltrombopag 50 mg/day for 3 weeks. At the end of these 3 weeks of treatment: platelet count higher than 100 x10e9/L and no spontaneous bleeding, end therapy. In the other cases, treatment with eltrombopag 75 mg/day for 3 additional weeks.
  Phase 2: Eltrombopag will be administered for 16 weeks. Eltrombopag will be initially given at 25 mg/day for 4 weeks. Every 4 weeks, the dosage will be modified as follows. (1) Bleeding score (WHO bleeding scale) 0-1 and platelet count between 30 and 100 x10e9/L: continue at the current dose; (2) Bleeding score 0-1 and platelet count higher than 100 x10e9/L: switch to the next lower dose; (3) Bleeding score 2-4 or platelet count lower than 30 x 10e9/L: switch to the next higher dose. The following dosages of eltrombopag are considered: 12.5 mg/day; 25 mg/day; 50 mg/day; 75 mg/day.
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag

SUMMARY:
Inherited thrombocytopenias (ITs) are a heterogeneous group of disorders characterized by a reduced number of blood platelets and a consequent bleeding tendency that ranges from mild to life-threatening. Thrombocytopenia is caused by genetic mutations and therefore is present throughout life and can be transmitted to the progeny. Some patients with severely reduced platelet count present spontaneous bleeding, which represents a major clinical problem: in fact, bleeding diathesis exposes these subjects to the risk of severe hemorrhages, affects their quality of life and often requires hospitalization and/or transfusions. Conversely, other patients with ITs have absent or mild spontaneous bleeding tendency. However, even these patients are at risk of major bleeding on the occasion of surgery or other invasive procedures. Therefore, the potential for hemorrhages on the occasion of invasive procedures represent a clinical problem for all patients affected by ITs.

Eltrombopag is a drug, available in tablets, which stimulates the production of platelets by the bone marrow. A previous study demonstrated that a short course of eltrombopag was effective in increasing platelet count in most patients with the MYH9-related disease (MYH9-RD), the most frequent form of IT. Eltrombopag was given for 3 to 6 weeks to 12 patients with MYH9-RD and platelet counts lower than 50 x10e9/L. Eleven patients responded to the drug and 8 of them obtained platelet counts higher than 100 x10e9/L or three times the baseline value. Remission of spontaneous bleeding was achieved by 8 of 10 patients and treatment was well tolerated in all the cases. Based on these findings, short-term eltrombopag courses have been successfully used for preparing for major surgery two patients with MYH9-RD and less than 20 x10e9 platelets/L.

The present study has two main objectives. - To verify if eltrombopag is effective in transiently increasing platelet count over 100 x 10e9/L and abolishing bleeding tendency in patients with different forms of IT.

To this end, eltrombopag will be given for 3-6 weeks to patients with different forms of IT. Eltrombopag will be administered at the dose of 50 mg/day for 3 weeks. After 3 weeks of treatment, the patients who will obtain a platelet count higher than 100 x10e9/L and complete remission of bleeding tendency will stop therapy. In the other cases, patients will be treated with eltrombopag at a higher dose (75 mg/day) for 3 additional weeks. This treatment schedule is called "Phase 1" of the study.

If the study will achieve this goal, short-term eltrombopag could be potentially used in the future to prepare these patients for surgery or other invasive procedures

- To verify if eltrombopag can be used to stably reduce spontaneous bleeding tendency for long periods of time in patients with clinically significant spontaneous hemorrhages.

To this end, patients with clinically significant spontaneous bleedings at baseline and who had their bleeding tendency reduced during the Phase 1 of the study without severe side effects, will be admitted to the "Phase 2" of the study.

During the Phase 2, patients will be treated with eltrombopag for 16 weeks. In order to determine the lowest dose of eltrombopag that is able to reduce or abolish their bleeding tendency, patients will start treatment with eltrombopag 25 mg/day for 4 weeks. Then, every 4 weeks, patients will be re-evaluated and the dosage of eltrombopag will be adjusted according to bleeding tendency and platelet count. The dosages of eltrombopag that can be used in the Phase 2 range from 12.5 to 75 mg/day.

Other objectives of the study are:

* to evaluate safety and tolerability of Eltrombopag in patients affected with ITs.
* to identify the dosages of Eltrombopag required for achieving the primary endpoints of Phases 1 and 2.
* to study the effects of Phase 2 treatment on patients' health-related quality of life (HR-QoL);
* to study the effects of treatment on some laboratory parameters related to platelet production and function.

All patients will be undergo a follow-up visit 30 days after completion of treatment.

Patients will be treated as outpatients. The evaluation of patients at enrollment and at each subsequent on-treatment and post-treatment visits includes: medical history; physical examination; evaluation of bleeding tendency according to WHO bleeding scale; CBC and differential; platelet count by phase-contrast microscopy; peripheral blood smear examination; plasma transaminases, bilirubin, and creatinine; urine analysis; ophthalmic assessment (only at some visits); measurement of serum thrombopoietin level; evaluation of HR-QoL (only at baseline and during Phase 2); evaluation of in vitro platelet aggregation in response to ADP, collagen and ristocetin whenever platelet count is over 100 x 10e9/L.

ELIGIBILITY:
Inclusion Criteria:

Phase 1:

Patients with the following forms of inherited thrombocytopenias will be considered for enrolment:

* MYH9-related disorders (OMIM 155100, 605249, 153640, 153650)
* Bernard-Soulier Syndrome (OMIM 231200) deriving from monoallelic mutations (at variance with biallelic classical BSS, monoallelic form does not present defective platelet function)
* Wiskott-Aldrich syndrome (OMIM 301000).
* X-linked thrombocytopenia (OMIM 313900).
* X-linked thrombocytopenia with thalassemia (OMIM 314050).
* Dyserythropoietic anemia with thrombocytopenia (OMIM 300367).
* ITGA2B/ITGB3-related thrombocytopenia (OMIM not available).
* ANKRD26-related thrombocytopenia (OMIM 188000).
* TUBB1-related thrombocytopenia (OMIM not available)
* ACTN1-related thrombocytopenia (OMIM not available)
* GFI1B-related thrombocytopenia (OMIM not available)
* CYCS-related thrombocytopenia (OMIM 612004)
* SLFN14-related thrombocytopenia (OMIM not available)

Patients will have to fulfill all the following criteria:

* Age ≥ 16 years and ≤ 70 years
* Average platelet count during the previous year less than 80 x109/L
* Written informed consent

Phase 2

Patients with clinically relevant chronic or recurrent bleedings at baseline (grade 2-4 of the WHO bleeding scale) who: (i) completed the phase 1 without severe side effects and (ii) obtained reduction or remission of bleeding by Eltrombopag administration.

Exclusion Criteria:

Phases 1 and 2

* Hypersensitivity to Eltrombopag or one of the excipients.
* History of thromboembolic events.
* Treatment with anti-platelet drugs or other drugs affecting platelet function and/or with anticoagulants.
* Concurrent diseases or conditions that significantly increase the risk of thromboembolic events.
* Moderate to severe liver failure (Child-Pugh score ≥ 5).
* Altered renal function as defined by creatinine ≥ 2 mg/dL
* Previous or concurrent clonal disorders of the myeloid series (acute myeloid leukemias and myelodysplastic syndromes).
* Females who are pregnant or nursing (a negative pregnancy test is required before enrolment of fertile women).
* Formal refusal of any recommendations for a safe contraception.
* Alcohol or drug addiction.
* Any other disease or condition that by the advice of the responsible physician would make the treatment dangerous for the patient or would make the patient ineligible for this study, including physical, psychiatric, social and behavioral problems.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
platelet count | 3 or 6 weeks (Phase 1)
  Phase 1: major response is defined by increase of platelet count over 100 x10e9/L and no bleeding tendency (grade 0 of the WHO bleeding scale) during the last week of treatment. Minor response is defined by a platelet at least two-fold increased with respect to baseline value without reaching the criteris for major response.
bleeding tendency according to the WHO bleeding scale | 3 or 6 weeks (Phase 1); 16 weeks (Phase 2)
  Phase 1: major response is defined by increase of platelet count over 100 x10e9/L and no bleeding tendency (grade 0 of the WHO bleeding scale) during the last week of treatment.
  Phase 2: Major response is defined as a complete remission of hemorrhages. Minor response is defined as a reduction of bleeding according to the WHO bleeding scale without reaching the criteria for major response.

SECONDARY OUTCOMES:
Daily dose of eltrombopag (in milligrams) required for achievement of the primary endpoints | 3 or 6 weeks (Phase 1); 16 weeks (Phase 2)
number and severity of adverse events as a measure of safety and tolerability. | 7 or 10 weeks (Phase 1); 20 weeks (Phase 2)
patients' health-related quality of life as a result of reduction of spontaneous bleeding tendency. | 20 weeks (Phase 2)

OTHER OUTCOMES:
serum thrombopoietin level | 7 or 10 weeks (Phase 1); 20 weeks (Phase 2)
  effect of treatment on serum thrombopoietin level
number of reticulated platelets | 7 or 10 weeks (Phase 1); 20 weeks (Phase 2)
  effect of treatment on number of reticulated platelets
in vitro platelet aggregation in response to different agonists as a measure of the function of platelets under eltrombopag treatment. | 7 or 10 weeks (Phase 1); 20 weeks (Phase 2)
In vitro platelet activation by flow cytometry analysis as a measure of the function of platelets under eltrombopag treatment. | 7 or 10 weeks (Phase 1); 20 weeks (Phase 2)

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Pecci, M.D., Principal Investigator — Unit of Internal Medicine 3, Department of Internal Medicine, IRCCS Policlinico San Matteo Foundation, Pavia, Italy
Locations (3):
- Italy (3):
  - Department of Internal Medicine, Hospital of Padova, Padua
  - Unit of Internal Medicine 3, IRCCS Policlinico San Matteo Foundation, Pavia
  - Section of Internal and Cardiovascular Medicine, Department of Medicine, University Hospital of Perugia, Perugia

REFERENCES:
- [Background] Balduini CL, Pecci A, Noris P. Diagnosis and management of inherited thrombocytopenias. Semin Thromb Hemost. 2013 Mar;39(2):161-71. doi: 10.1055/s-0032-1333540. Epub 2013 Feb 8. PMID 23397552
- [Background] Pecci A. Pathogenesis and management of inherited thrombocytopenias: rationale for the use of thrombopoietin-receptor agonists. Int J Hematol. 2013 Jul;98(1):34-47. doi: 10.1007/s12185-013-1351-7. Epub 2013 May 1. PMID 23636669
- [Background] Pecci A, Gresele P, Klersy C, Savoia A, Noris P, Fierro T, Bozzi V, Mezzasoma AM, Melazzini F, Balduini CL. Eltrombopag for the treatment of the inherited thrombocytopenia deriving from MYH9 mutations. Blood. 2010 Dec 23;116(26):5832-7. doi: 10.1182/blood-2010-08-304725. Epub 2010 Sep 15. PMID 20844233
- [Background] Pecci A, Barozzi S, d'Amico S, Balduini CL. Short-term eltrombopag for surgical preparation of a patient with inherited thrombocytopenia deriving from MYH9 mutation. Thromb Haemost. 2012 Jun;107(6):1188-9. doi: 10.1160/TH12-01-0005. Epub 2012 Mar 8. No abstract available. PMID 22398565
- [Background] Favier R, Feriel J, Favier M, Denoyelle F, Martignetti JA. First successful use of eltrombopag before surgery in a child with MYH9-related thrombocytopenia. Pediatrics. 2013 Sep;132(3):e793-5. doi: 10.1542/peds.2012-3807. Epub 2013 Aug 12. PMID 23940247
- [Derived] Zaninetti C, Gresele P, Bertomoro A, Klersy C, De Candia E, Veneri D, Barozzi S, Fierro T, Alberelli MA, Musella V, Noris P, Fabris F, Balduini CL, Pecci A. Eltrombopag for the treatment of inherited thrombocytopenias: a phase II clinical trial. Haematologica. 2020 Mar;105(3):820-828. doi: 10.3324/haematol.2019.223966. Epub 2019 Jul 4. PMID 31273088